# Safety and Feasibility Testing of a Smaller Network Version of AIDANET

Running Title: Smaller Network Pilot

NCT06633965

Version Number:

v1.3 25-Oct-2024



# **KEY ROLES**

| | Name, Degree | Institution Name |
|---|---|---|
| Principal Investigator, IDE<br>Chair | Marc D. Breton, PhD | University of Virginia Center for Diabetes Technology |
| Protocol Chair | Sue A. Brown, MD | University of Virginia Center for Diabetes Technology |
| Study Physician | Mark D. DeBoer, MD | University of Virginia Center for Diabetes Technology |

MiniNET\_25-Oct-2024 



# PROTOCOL VERSION HISTORY

| Version<br>Number | Author(s) | Approver | Effective Date | Revision Description |
|---|---|---|---|---|
| 1.0 | Sue Brown | Sue Brown,<br>Mark DeBoer | 11-Sep-2024 | Original Protocol |
| 1.1 | Mary Oliveri | Sue Brown,<br>Mark DeBoer | 24-Sep-2024 | FDA Modifications: • Modified Glycemic Treatment Guidelines (section 7.6.1) • Modified Stopping Criteria (section 12.9.1) |
| 1.2 | Mark DeBoer | Sue Brown,<br>Mark DeBoer | 25-Sep-2024 | FDA Modifications: • Modified Glycemic Treatment Guidelines (section 7.6.1) |
| 1.3 | Mary Oliveri | Mary Oliveri | 25-Oct-2024 | Study Team Modifications: • Added definition of AIDANET acronym (section 1.1) • Removed activity tracker (section 4.3) IRB Modifications: • Removed reference to assent (section 3.3) • Removed pregnancy test at hotel visit (section 7.3) |

MiniNET\_25-Oct-2024 



#### SITE PRINCIPAL INVESTIGATOR STATEMENT OF COMPLIANCE

Protocol Title: Safety and Feasibility Testing of a Smaller Network Version of AIDANET

Running Title: Smaller Network Pilot

Protocol Version/Date: v1.3/25-Oct-2024

I have read the protocol specified above. In my formal capacity as a Site Principal Investigator, my duties include ensuring the safety of the study participants enrolled under my supervision. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site.

This trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP) and as required by the following: United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

As the Principal Investigator, I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), or other approved Ethics Committee, except where necessary to eliminate an immediate hazard(s) to the trial participants.

All key personnel (all individuals responsible for the design and conduct of this trial) have completed Human Participants Protection Training and Good Clinical Practice Training. Further, I agree to ensure that all staff members involved in the conduct of this study are informed about their obligations in meeting the above commitments.

| Investigator's Signature | Date: | / | / |
|-----------------------------------|-------|---|---|
| Investigator's Name: | | | |
| Site Name: University of Virginia | | | |

MiniNET 25-Oct-2024 



# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|--------------------------------------------------------------|
| ADA | American Diabetes Association |
| AE | Adverse Event |
| AID | Automated insulin delivery |
| AIDANET | Automated insulin delivery as Adaptive Network |
| AP | Artificial pancreas |
| AUC | Area Under the Curve |
| AYA | Adolescent and Young Adult |
| BDC | Barbara Davis Center |
| BG | Blood Glucose (as assessed by a blood glucose meter) |
| BGM | Blood glucose meter |
| CGM | Continuous glucose monitor |
| CSII | Continuous subcutaneous insulin infusion |
| DiAs | Diabetes Assistant |
| DKA | Diabetic Ketoacidosis |
| FCL | Fully closed loop |
| HbA1c | Hemoglobin A1c |
| HCL | Hybrid closed loop |
| JDRF | Juvenile Diabetes Research Foundation |
| MDI | Multiple daily injections |
| NAP | Neural network artificial pancreas |
| SAE | Severe Adverse Event |
| SG | Sensor Glucose (as assessed by a continuous glucose monitor) |
| SH | Severe Hypoglycemia |
| T1D | Type 1 diabetes |
| TAR | Time above range |
| TBR | Time below range |
| TIR | Time in range 70-180 mg/dL |

MiniNET\_25-Oct-2024 



# PROTOCOL SUMMARY

| Participant Area | Description |
|---|---|
| Title | Safety and Feasibility Testing of a Smaller Network Version of AIDANET |
| Investigational<br>Device | AIDANET algorithm as smaller network version with DiAs phone, Tandem t:AP insulin pumps, and Dexcom CGM |
| Objectives | The primary objective of the project is to demonstrate feasibility and safety of the Automated Insulin Delivery as Adaptive NETwork (AIDANET) system run in a new smaller network version, used in full closed loop (FCL) by adults with T1D. |
| Study Design | Randomized crossover, device safety/feasibility supervised house/hotel with transition to home use, interventional trial of AIDANET |
| Number of Sites | 1 |
| Endpoint | The primary metric for analysis will be change in mean CGM between the week of the control usual-care period and the one-week Remote Monitored At-Home Full Closed Loop period using AIDANET. |
| Population | <ul> <li>Key Inclusion Criteria</li> <li>Age 18-60 years at time of consent.</li> <li>Clinical diagnosis of T1D, based on investigator assessment, of at least 1 year duration.</li> </ul> |
| Sample Size | Complete 6 participants |
| Treatment Groups | Randomized Crossover: Participants will be randomized 1:1 to either conduct the control period before use of the AIDANET system (Group A) or after use of the AIDANET system (Group B). |
| Participant Duration | Approximately 3 weeks: approximately 1 week of usual care, 3 days/2 nights house/hotel in FCL, and 1 week At Home Remote Monitored FCL. |
| Protocol<br>Overview/Synopsis | We will enroll up to 12 participants with a plan to complete 6 participants. The study will be performed for about 36 hours at a local hotel/rental. Following the house/hotel session, participants will undergo a 7 day/6-night Remote Monitored At-Home use session. We will also conduct a one-week control period gathering data on glycemic control and insulin administration with the participants usual care therapy. Participants will be randomized 1:1, to either Group A (control period prior to AIDANET use) or Group B (control period after AIDANET use). |

MiniNET\_25-Oct-2024 

## TABLE 1. SCHEDULE OF STUDY VISITS AND PROCEDURES

| | Screening | Randomization | Usual Care<br>Data<br>Collection | Pre-Hotel<br>Check In | Hotel<br>Admission<br>with FCL | FCL<br>Equipment<br>Training | 1-week<br>at-home<br>FCL | Post Study<br>Check-In |
|---|---|---|---|---|---|---|---|---|
| Location | CV/R/Ph | CV/R/Ph | Home x 1<br>week | R/Ph | House/<br>Hotel | House/<br>Hotel | Home x 1<br>week | Home |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| Timeframe (days) | 1 | 2 | 3-10 | 11 | 12-14 | 12 | 14-21 | 22 |
| Informed Consent | X | | | | | | | |
| Eligibility<br>Assessment | X | | | | | | | |
| Medical History | X | | | | | | | |
| HbA1c | X | | | | | | | |
| Pregnancy Test (if applicable) | X | | | | | | | |
| Blood Testing:<br>BMP, Liver<br>Functioning,<br>Hematocrit, TSH<br>(if requested by<br>MD) | X | | | | | | | |
| Physical Exam<br>(H&P within 6<br>months permitted<br>as substitute) | X | | | | | | | |
| Vital Signs (including height/weight) (self-reported values permitted) | X | | | | X | | | |

MiniNET\_25-Oct-2024 

| Demographic Data<br>Survey (if<br>eligibility is met) | X | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Randomization | | X | | | | | | |
| Study Equipment<br>Training | | | | | | X | | |
| CGM Use | | | X | X | X | X | X | |
| Fully Closed Loop<br>(FCL) Use (e.g.<br>AIDANET, DiAs,<br>CGM) | | | | | X | Х | X | |
| Questionnaires | | | | | X | | X | |
| Concomitant<br>Medication Review | X | | | | X | | | |
| Review diabetes<br>management and<br>AEs | | | X | X | X | X | X | X |

CV = Clinic Visit; R=Remote Visit; Ph=Phone which includes text messages and emails

MiniNET\_25-Oct-2024 

**Table 2. Metric Capture Timeline** 

| | Enrollment | 1-Week<br>Usual Care | Hotel FCL | 1-Week at-<br>home FCL |
|---|---|---|---|---|
| Visit | 1 | 3 | 5 | 7 |
| Demographic Data | X | | | |
| HbA1c | X | | | |
| CGM Data | | | | |
| Mean CGM | | X | X | X |
| GMI | | X | X | X |
| TIR 70-180 mg/dL | | X | X | X |
| CGM StDev | | X | X | X |
| CGM CV | | X | X | X |
| CGM%<54 mg/dL | | X | X | X |
| CGM%<70 mg/dL | | X | X | X |
| CGM%>180 mg/dL | | X | X | X |
| CGM%>250 mg/dL | | X | X | X |
| Time in Automation | | | X | X |
| Total Daily Insulin Dose | | X | X | X |
| Number of Boluses per Day | | X | X | |
| Exercise: CGM %<70 mg/dL | | | X | |
| Unannounced Meals: % CGM>250 mg/dL | | | Х | |
| Inspire Questionnaire | | | X | X |
| Technology Expectations Survey | | | X | X |

MiniNET\_25-Oct-2024 

| 1 | Table of Contents | |
|----|---------------------------------------------------|----|
| 2 | Chapter 1: Background | 14 |
| 3 | 1.1 Introduction | 14 |
| 4 | 1.2 Study Objective | |
| 5 | 1.3 Specific Aims and Hypotheses | 15 |
| 6 | Chapter 2: Study Synopsis | 16 |
| 7 | 2.1 Study Design | 16 |
| 8 | 2.2 Study Hardware/Software | 16 |
| 9 | 2.3 Timing of Device Use | 16 |
| 10 | 2.4 Meal and Exercise Testing | 17 |
| 11 | 2.5 Study Devices Download | |
| 12 | 2.6 Study System Issues | 18 |
| 13 | Chapter 3: Study Screening | 19 |
| 14 | 3.1 Clinical Site | 19 |
| 15 | 3.2 Participant Recruitment and Enrollment | 19 |
| 16 | 3.3 Informed Consent and Authorization Procedures | 19 |
| 17 | 3.4 Participant Inclusion Criteria | 19 |
| 18 | 3.5 Participant Exclusion Criteria | 20 |
| 19 | 3.6 Screening Procedures | 21 |
| 20 | 3.7 Screen Failures | 22 |
| 21 | 3.8 Personal Equipment Downloads | 23 |
| 22 | 3.9 Questionnaire | 23 |
| 23 | 3.10 Other Considerations | 23 |
| 24 | Chapter 4: Study Devices & Training | 24 |
| 25 | 4.1 Insulin Pump | 24 |
| 26 | 4.2 Continuous Glucose Monitor | 25 |
| 27 | 4.3 Blood Glucose Meter and Strips | 26 |
| 28 | 4.4 Ketone Meter and Strips | 26 |
| 29 | 4.5 Study Devices Accountability Procedures | 26 |

| Chapter 5: Randomization | <br>27 |
|-----------------------------------------------------------------|--------|
| Chapter 6: Usual Care Control Period | 28 |
| 6.1 Usual Care Control Period | 28 |
| 6.2 Pre-Hotel Check-In Visit | 28 |
| Chapter 7: Supervised Hotel Fully Closed Loop Period | 29 |
| 7.1 Hotel Session | 29 |
| 7.2 Qualifications and Role of the Staff | 29 |
| 7.3 Hotel Session Check-In | 29 |
| 7.4 Study Meals | 30 |
| 7.5 Hotel Session Activities | 30 |
| 7.6 Glycemic Treatment Guidelines | 30 |
| 7.7 FCL Equipment Training | 31 |
| 7.8 Hotel Session Discharge | 31 |
| 7.9 Other Issues | 32 |
| Chapter 8: Remote Monitored At-Home Fully Closed Loop Period | 33 |
| 8.1 At Home Participant Plan | 33 |
| 8.2 Remote Monitoring. | 33 |
| 8.3 Questionnaires | 33 |
| 8.4 Post-Study Check-In | 34 |
| 8.5 Early Termination Visit (If Applicable) | 34 |
| 8.6 Unscheduled Visits | 34 |
| Chapter 9: Medical Monitor Safety Review | 35 |
| Chapter 10: Testing Procedures | 36 |
| 10.1 Laboratory and Point of Care Testing | 36 |
| 10.2 Questionnaires | 36 |
| Chapter 11: Risks Associated with the Clinical Trial | 38 |
| 11.1 Potential Risks and Benefits of the Investigational Device | 38 |
| 11.2 General Considerations | 41 |

| 58 | Chapter 12: Adverse Events, Device Issues, and Stopping Rules | 43 |
|----|---------------------------------------------------------------|----|
| 59 | 12.1 Definitions | 43 |
| 60 | 12.2 Reportable Events | 44 |
| 61 | 12.3 Relationship of Adverse Event to Study Device | 45 |
| 62 | 12.4 Intensity of Adverse Event | 45 |
| 63 | 12.5 Coding of Adverse Events | 46 |
| 64 | 12.6 Outcome of Adverse Events | 46 |
| 65 | 12.7 Reportable Device Issues | 47 |
| 66 | 12.8 Timing of Event Reporting | 47 |
| 67 | 12.9 Stopping Criteria | 48 |
| 68 | 12.10 Independent Safety Oversight | 48 |
| 69 | 12.11 Definition of a Data Breach | 49 |
| 70 | Chapter 13: Miscellaneous Considerations | 50 |
| 71 | 13.1 Prohibited Medications, Treatments, and Procedures | 50 |
| 72 | 13.2 Participant Withdrawal | 50 |
| 73 | 13.3 Confidentiality | 50 |
| 74 | 13.4 Lost to Follow Up | 50 |
| 75 | Chapter 14: Statistical Consideration | 51 |
| 76 | 14.1 Design and Randomization | 51 |
| 77 | 14.2 Sample Size | 51 |
| 78 | 14.3 Outcome Measures | 52 |
| 79 | 14.4 Safety Analyses | 53 |
| 80 | 14.5 Baseline Descriptive Statistics | 53 |
| 81 | 14.6 Device Issues | 54 |
| 82 | Chapter 15: Data Collection and Monitoring | 55 |
| 83 | 15.1 Case Report Forms and Device Data | 55 |
| 84 | 15.2 Study Records Retention | 55 |
| 85 | 15.3 Protocol Deviations | 55 |
| 86 | Chapter 16: Ethics/Protection of Human Participants | 56 |

| 87 | 16.1 Ethics Standard | 56 |
|----|-------------------------------------------|----|
| 88 | 16.2 Institutional Review Boards | 56 |
| 89 | 16.3 Informed Consent Process | 56 |
| 90 | 16.4 Participant and Data Confidentiality | 57 |
| 91 | Chapter 17: References | 58 |
| 92 | | |
| 93 | | |

MiniNET\_25-Oct-2024 

# **Chapter 1: Background**

## 1.1 Introduction

94

95

121

122

123

124125

126

127128

96 A major impediment to maintaining blood glucose (BG) control in Type 1 diabetes (T1D) is missed meal boluses, which has been associated with significantly higher HbA1c levels. While the 97 advent of the artificial pancreas (AP) offers promise of safe reductions in HbA1c, our research 98 group previously found that current AP systems only partly compensate for missed prandial 99 insulin.<sup>2</sup> We thus designed a new system called Automated Insulin Delivery Adaptive NETwork, 100 101 or AIDANET, to be fully automated, utilizing a Bolus Priming System (BPS) that recognizes meal ingestion and delivers a quick priming dose of insulin prior to extreme blood sugar excursions. 102 103 When used as a fully automated closed loop (FCL) system (without any meal announcements to the controller), this system improves glucose time-in-target range (TIR) 70-180 mg/dL compared 104 to a current commercially available system (Control-IQ). We subsequently incorporated this 105 106 system in a neural net and found this to function as well as the previous model-predictive control algorithm. However, the long-term utility of such a system would have to be via use on an insulin 107 108 pump, requiring a refined "smaller" code set to be able to run on internal pump software.

- 109 We have thus formulated a version of AIDANET that has a smaller coding footprint. The goal of the current project is to assess whether this "smaller" version of AIDANET continues to provide 110 111 safe and effective glycemia management as seen in prior formulations. The current study is a 112 randomized cross-over study comparing participants' usual care with one week at home on 113 AIDANET. The week of control at home will follow a two-night hotel stay when participants will be taught how to operate the new system during the at-home portion of the study. The comparator 114 usual care week will be randomly assigned to being before time on AIDANET (i.e., prior to the 115 116 hotel stay) or after (i.e. time after the one-week home portion).
- For the majority of time on AIDANET, participants will not announce meal ingestion to the system—using the system as an FCL system. However, the system is designed to also be able to be used as a hybrid system with carbohydrate announcement. Thus, as further assessment of the system, we will instruct participants to use the system as follows:
  - For one of the dinners in the hotel participants will bolus for carbohydrate content of their meal, using their usual insulin-to-carbohydrate ratio (while the other dinner in the hotel will be fully FCL).
  - For one full day while at home participants will bolus for carbohydrates for all ingestions (using their usual insulin-to-carbohydrate ratio).
  - For another full day at home, participants will merely announce to the system each time they begin to eat a meal or snack; this will induce the system to deliver a rapid BPS dose (e.g. 10% of total daily insulin).

We hypothesize that performances of this smaller version of AIDANET will provide safe and effective care when used as FCL (with the exception of the hybrid use as just described). We expect

MiniNET 25-Oct-2024 

- that this will constitute an important step toward having an AID system that has potential to be
- used embedded in insulin pumps.
- 133 **1.2 Study Objective**
- 134 This study aims to demonstrate the safety and feasibility of the Automated insulin delivery as
- Adaptive NETwork (AIDANET) system in a smaller software version, used as FCL. This study
- will also assess differences in glycemia outcomes on assigned days when the participant 1) enters
- total carbohydrate amount and 2) announces when food is started to be consumed.
- 138 1.3 Specific Aims and Hypotheses
- 139 Aim 1: To evaluate the performance (safety, efficacy) of the smaller version of AIDANET used
- as FCL.
- 141 **Hypothesis:** FCL use will provide as good or better mean CGM value and glucose TIR during 1
- week of at-home use as compared to 1 week of standard care sensor data.
- 143 Aim 2: To evaluate the safety and efficacy of the smaller version of AIDANET during days where
- participants are assigned to 1) use usual insulin-to-carbohydrate ratio and 2) use meal
- announcement alone (triggering BPS).
- 146 **Hypothesis:** The AIDANET system will yield improved mean CGM glucose and TIR on days
- 147 when meals are announced, both using insulin-to-carbohydrate ratio and simple meal
- 148 announcement.

MiniNET 25-Oct-2024 

# **Chapter 2: Study Synopsis**

## 2.1 Study Design

This study assesses adults with T1D on the AIDANET system during a 2-night house/hotel stay and during 1 week at home (Figure 1). Participants will use the system as FCL with the exception of using their insulin-to-carbohydrate ratio as usual during 1 dinner in the house/hotel and 1 day at home and announcing eating initiation for 1 day at home. We will aim to complete a total of 6 participants. We will also conduct an approximately 1-week control period gathering data on glycemic control and insulin administration with the participants' usual care therapy. Participants will be randomized 1:1 to either Group A (control period prior to AIDANET use) or Group B (control period after AIDANET use).



• Figure 1: Device Use Timeline

#### 2.2 Study Hardware/Software

The study will involve testing a new AID system designed to enable full closed loop control and consisting of the following elements: the diabetes assistant (DiAs) prototyping platform, connected to a Tandem t:AP research insulin pump and a Dexcom G6 CGM, and implementing a new "smaller" coding version of the University of Virginia (UVA) AIDANET algorithm. Upon arrival at the hotel, participants will be taught how to use the Tandem t:AP pump as well as the DiAs system, including stopping the system.

## 2.3 Timing of Device Use

*One-Week Control Period*: All participants will collect approximately one week of usual care data to serve as control data for cross-over testing as outlined in Section 6.1. During the control period, participants may use an insulin pump either in manual or automated mode that is capable of being downloaded. Participants will be randomized 1:1 to either conduct the control period before use of the AIDANET system (Group A) or after use of the AIDANET system (Group B).

MiniNET 25-Oct-2024 

- 174 *Hotel Period*: Participants will arrive at the hotel prior to dinner on the afternoon of Day 1. They
- will be connected to the Tandem t:AP pump, which will be connected to the DiAs platform. A
- Dexcom G6 CGM may be placed on Day 1 or by the participant prior to Day 1 and will also be
- 177 connected to the DiAs platform. The system will be started in the afternoon/evening with
- 178 AIDANET enabled prior to dinner on Day 1. Participants will be taught how to use the DiAs in
- this configuration. The t:AP pump will be programmed with back up parameters determined by
- the study investigator(s). Once started, the participants will have their glucose values managed
- through use of this system during the hotel and Remote Monitored At-Home periods.
- 182 Remote Monitored At-Home Period: Participants will continue to use the Tandem t:AP pump,
- DiAs platform running the AIDANET smaller network system, and Dexcom G6 CGM for glucose
- 184 control for 7 days/6 nights during this period. At the end of the Remote Monitored At-Home
- period, participants will return to their usual diabetes therapy.

## 2.4 Meal and Exercise Testing

186

187

188

189

190

191

192

193

194

195

196

197

198

199

200

201202

203204

205

206

207

208

209

## 2.4.1 Meal Testing

During the supervised house/hotel period, participants will be instructed to eat approximately 3 unannounced meals per full day, with the exception of using their usual insulin-to-carbohydrate ratio with dinner one of the 2 nights. The time of completion for these meals will be recorded by study staff. The % CGM>250 mg/dL for the 4 hours after each meal will be recorded and specifically analyzed along with the CGM area under the curve (AUC) for the post-meal 4-hour period. Participants will be instructed to freely eat unannounced meals during the remotemonitored at-home stage but will not be required to record the timing of the meals. The exception is they will be instructed for 1 full day (from waking through bedtime) to announce usual insulinto-carbohydrate for all ingestions and for another full day to announce when they begin to eat. Participants will be educated to consume their usual diet during both the at-home control period and the Remote Monitored At-Home FCL period.

## 2.4.2 Exercise Testing

During the supervised hotel period, participants will engage in mild activity (a walk of approximately 30 minutes) on Day 2. Study staff will set a Temporary Control Rate (TCR) of approximately 50-100% starting up to approximately one hour prior to exercise for approximately 2 hours, actual TCR settings will be tailored to an individual person. Study staff will record the duration, approximate intensity (low, moderate, or high intensity), the TBR <70 mg/dL, TBR <54 mg/dL, and any episodes of Severe Hypoglycemia (SH) during the walk and in the 2 hours after the exercise challenges. Participants will be provided with an exercise monitor (e.g., Fitbit) for use during the control and FCL periods. Participants will be allowed to practice their usual exercise routine during the control and remote-monitored at-home FCL periods with use of the TCR as needed. They will not be required to record exercise events during these periods.

MiniNET 25-Oct-2024 

# 2.5 Study Devices Download Data from the study devices will be captured in real-time by the remote monitoring server for the

- 212 DiAs system. In addition, study devices will be downloaded at the end of the Remote-Monitored
- 213 At-Home FCL period.
- 214 **2.6 Study System Issues**
- 215 If the CGM signal becomes unavailable for more than 20 minutes consecutively, closed loop will
- 216 not operate to automatically adjust insulin delivery. If the CGM is not connected, the system will
- revert to the usual open loop function of the pump and deliver insulin with the pre-programmed
- dosing parameters. Resumption of closed-loop control will occur automatically once the CGM
- signal is again available.
- 220 If the DiAs system is unable to maintain connectivity with the Tandem t:AP pump, the pump will
- automatically revert to the pre-programmed dosing parameters after 30 minutes without any need
- for interaction from the user.

MiniNET 25-Oct-2024 

# 223 Chapter 3: Study Screening

- 224 **VISIT 1**
- 225 3.1 Clinical Site
- The study will be performed at the University of Virginia. Screening procedures will be performed
- either virtually or on site, at a clinical research unit, or at the hotel.
- 228 **3.2** Participant Recruitment and Enrollment
- We will enroll up to 12 participants who have been diagnosed with type 1 diabetes for at least one
- 230 year. This enrollment number accounts for dropouts or screen failures that may occur. The goal is
- 231 to complete a total of approximately 6 participants.
- 232 **3.3** Informed Consent and Authorization Procedures
- 233 Before consent has been obtained, participants will be asked inclusion/exclusion criteria questions
- 234 during pre-screening to determine study eligibility. Before completing any procedures or
- collecting any data that are not part of usual care, written informed consent will be obtained.
- Potential eligibility may be assessed as part of routine care examination.
- 237 A participant is considered enrolled when the informed consent forms have been signed by the
- participant and the study team.
- 239 Consenting procedures and documentation are defined in section 16.3.
- 240 After informed consent has been signed, a potential participant will be evaluated for study
- 241 eligibility through review of medical history, performance of physical exam by a licensed health
- care professional, and other testing as needed per the I/E criteria.
- 243 **3.4 Participant Inclusion Criteria**
- 244 The participants must meet all of the following inclusion criteria in order to be eligible to
- 245 participate in the study.

251

- 1. Age  $\geq$ 18.0 and  $\leq$ 60 years old at time of consent
- 247 2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
- 249 3. Currently using insulin pump for at least three months; Any pump, either open loop or hybrid closed loop may be used.
  - 4. Currently using insulin for at least six months.
- 5. Willingness to switch to use a commercially approved personal insulin (e.g., lispro or aspart, or biosimilar approved products) within the study pump as directed by the study team.

MiniNET 25-Oct-2024 

256

257

258

259260

261262

263

264

265

266

267

268

269

270

271

272

273

274

275

276

277

278

279

286

289

- 6. Currently using a Dexcom G6 or G7 CGM.
  - 7. Has one or more supportive companions knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff that either lives with participant or located within approximately 30 minutes of participant and able to locate participant in the event of an emergency.
  - 8. Participant not currently known to be pregnant or breastfeeding.
  - 9. If participant capable of becoming pregnant, must agree to use a form of contraception to prevent pregnancy while a participant in the study (e.g. hormonal contraception, abstinence from heterosexual intercourse). A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
  - 10. Willingness to use the study FCL system (CGM, pump, and phone) during the relevant study period.
  - 11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
  - 12. Willingness to participate in all study procedures including the house/hotel session, exercise challenges (e.g., one hour per day during hotel), and to consume approximately 3 unannounced meals per day during the relevant portion of the supervised hotel session.
  - 13. Access to internet at home and willingness to upload data during the study as needed.
  - 14. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
  - 15. Participant is proficient in reading and writing English.

## 3.5 Participant Exclusion Criteria

- The participant must not have any exclusion criteria in order to be eligible to participate in the study.
- 282 1. Plans to start a new non-insulin glucose-lowering agent (e.g., GLP-1 receptor agonists, Symlin, DPP-4 inhibitors, sulfonylureas). Participants may be on a stable dose of such an agent for at least the past month.
- 285 2. Current use of an SGLT-2 or SGLT-1/2 inhibitor due to risk of euglycemic DKA.
  - 3. Hemophilia or any other bleeding disorder.
- 4. History of severe hypoglycemic events with seizure or loss of consciousness in the last 12
   months.
  - 5. History of DKA event in the last 12 months.
- 290 6. History of chronic renal disease (Stage 4 or unstable Stage 3b per investigator judgment) 291 or currently on peritoneal or hemodialysis.

MiniNET 25-Oct-2024 

323

324

325

326

327

328

329

g. History of seizures

h. Loss of consciousness

4. Basal rates or basal insulin dosing

5. Carbohydrate ratios

8. Average daily insulin

7. Target glucose

6. Insulin sensitivity factors

292 7. History of adrenal insufficiency. 293 8. Currently being treated for a seizure disorder. 9. Hypothyroidism or hyperthyroidism that is not adequately treated. 294 10. Coronary artery disease or other heart condition that would prevent participation in 295 296 moderate intensity exercise. 297 11. Use of oral or injectable steroids at the time of enrollment or within the last 4 weeks. 12. Planned surgery during the study period. 298 299 13. Known ongoing adhesive intolerance that is not well managed. 14. A condition, which in the opinion of the investigator or designee, would put the 300 301 participant or study at risk. 302 15. Participation in another interventional trial at the time of enrollment. 303 16. Participant with a direct supervisor involved in the conduct of the trial. 304 3.6 Screening Procedures 305 The participant will be evaluated for study inclusion and exclusion eligibility after the informed 306 consent forms have been signed by the participant and the study team. Screening procedures will 307 last approximately 1-2 hours. The visit may occur in-person or remotely by HIPAA compliant 308 video communication (e.g., Zoom, Webex) The following procedures may be performed/data 309 collected/eligibility criteria checked and documented: 310 1. Inclusion and Exclusion criteria assessed 311 2. Demographics, including: 312 a. Date of birth 313 b. Gender 314 c. Race d. Ethnicity 315 316 3. Medical History, including diabetes history 317 a. Duration of disease (number of years) 318 b. History of pump use 319 c. History of CGM use 320 d. Current treatment 321 e. Severe hypoglycemia history 322 f. DKA history

MiniNET 25-Oct-2024 

| 330 | 9. Surgical history |
|---|---|
| 331 | 10. Allergies |
| 332 | 11. Concomitant medications |
| 333 | 12. Physical Examination – A historical history and physical report within 6 months of |
| 334 | screening appointments may be used but is not required for eligibility. If vitals are not |
| 335 | available, may include self-reported values of all available vitals. |
| 336 | a. Weight |
| 337 | b. Height |
| 338 | c. Blood pressure |
| 339 | d. Temperature |
| 340 | e. Heart Rate |
| 341 | 13. Screening Labs |
| 342 | a. HbA1c point of care or laboratory; may use an HbA1c if obtained in the past month. |
| 343 | b. Urine or serum pregnancy test for all women of childbearing potential (this test can |
| 344 | be done remotely with results sent to the study team) |
| 345<br>346<br>347<br>348<br>349 | A physical exam documented in the prior 12 months can suffice for the physical exam but will not serve as an exclusion criterion if not available. Participants may self-report height, weight, blood pressure, temperature, and heart rate; or these may be obtained by study staff at the enrollment visit. An HbA1c value obtained in the previous one month may serve for the enrollment HbA1c value. |
| 350<br>351<br>352<br>353<br>354 | If needed based on medical history, investigators may include baseline chemistry panel, liver function tests, hematocrit, and thyroid stimulating hormone (lab results within one year of screening appointment may be used). Any labs required may be obtained at a local laboratory (e.g., LabCorp, Quest) convenient to the participant. The study physician or physician designee will have the discretion to repeat screening tests if applicable. |
| 355 | 3.7 Screen Failures |
| 356<br>357 | If an exclusionary condition is identified, the study participant will be excluded from participation with follow up and referral to their primary care physician as needed. |
| 358<br>359<br>360 | If the study participant is pregnant, the study physician will discuss the results of the blood test with the participant and the participant will be asked to seek confirmation of the test and the appropriate medical care. |
| 361<br>362 | Participants may be re-screened if their clinical situation changes as determined by the study physician. |

MiniNET\_25-Oct-2024 

## 363 3.8 Personal Equipment Downloads Up to 6 months of historical data from the participant's personal insulin pump, glucometer, or 364 continuous glucose monitor may be downloaded or recorded. Data will be obtained from the 365 366 participant's personal insulin pump, glucometer and CGM. This data may be obtained through the 367 commercial applications (e.g., t:connect, Tidepool, and Dexcom). 368 3.9 Questionnaire 369 Participants will be asked to complete the Demographic Data Survey, as described in section 9.2, 370 once eligibility has been met. 371 3.10 Other Considerations 372 This study is not meant to find out if the participant has any other disease or problem. The study leaders will alert the participant if any of the research results are important to the participant's 373 374 health during the study. The participant may have a copy of the screening tests to discuss with the personal physician. If blood tests are completed, any blood left over will be thrown away. It will 375 not be stored for any future testing. 376

MiniNET\_25-Oct-2024 

# **Chapter 4: Study Devices & Training**

- 378 The study system is designed to enable full closed loop control and consisting of the following
- elements: the diabetes assistant (DiAs) prototyping platform (smart phone), connected to a Tandem
- 380 t:AP research insulin pump and a Dexcom G6 CGM, and implementing a new "smaller" coding
- version of the University of Virginia (UVA) AIDANET algorithm.

## 4.1 Insulin Pump

377

382

383

397

398

399

400

401

402

403

404

## 4.1.1 Equipment Description.

- A study insulin pump will be provided to all participants at the training session. The participants
- will be trained in the basic functionality (e.g., bolus menu and infusion set change menu) for the
- 386 study pump. For the Tandem pumps a training checklist is available on-line with relevant sections
- applicable to the study pump will be covered.
- 388 The t:AP research CSII pump will be programmed with the participants' usual pump parameters
- 389 (basal insulin rate, insulin to carbohydrate ratio, and insulin correction factor) as determined by
- 390 the study physician at the onset of the hotel phase. These parameters serve as backup-only settings
- 391 for the system in open loop mode, and do not determine behavior of the AIDANET algorithm. The
- 392 bolus priming system (BPS) profile determines the maximum fraction of total daily insulin (TDI)
- that can be injected by the BPS depending on the time of day (e.g., 8% between 06:00 and 10:00).
- 394 The BPS profile is a setting on DiAs which can be modified by the provider to impact performance
- of the AIDANET algorithm. The study physician may alter the BPS profile during the hotel and
- 396 at-home portions of the study to optimize participant safety with the experimental system.

## 4.1.2 Equipment Training

- Training on the DiAs and study pump may begin at the hotel after the AIDANET system has been put in place. The purpose of this training is to introduce the study system to the participant. Insulin parameters will be determined by the investigator(s) and programmed into their study insulin pump and confirmed by two research staff. Participants will then switch to the study insulin pump. The participant's personal pump will be removed. The investigator may elect to use an existing personal pump infusion site at their discretion at the start of the study. The participant will be instructed on charging the pump, menu navigation, bolus procedures, and infusion site changes.
- Data-driven optimization of pump settings can occur at any time prior to the hotel session,
- 406 particularly if the participant contacts the study physician due to concerns about their pump
- settings due to recurring hypo- or hyperglycemia. During closed loop testing, study investigators
- 408 may change pump settings as needed to optimize participant safety with the experimental system.

MiniNET 25-Oct-2024 

409

410

415

## **4.2 Continuous Glucose Monitor**

## **4.2.1 Equipment Description**

- The study CGM will include the Dexcom G6 transmitter and sensor. Participants may elect to wear
- their personal Dexcom G6 CGM equipment throughout the study period. If currently wear a G7
- 413 CGM model, the participant will be provided with G6 CGM supplies. These sensors may be worn
- for up to 10 days of continuous wear. The G6 transmitter may be worn for 3 months.

## 4.2.2 CGM Training

- 416 A study CGM will be provided to all participants at the training session which is expected to occur
- prior to the hotel session or prior to the usual care period based on the current use of CGM and
- 418 randomization. Participants using the Dexcom G6 may continue their personal CGM during the
- study session. The participants will be provided with CGM equipment and instructed to use CGM
- on a daily basis. If the participant has prior use of the G6, retraining will be specific to the
- individual. The study team may elect to have less frequent CGM users watch the Dexcom online
- 422 training videos (https://www.dexcom.com/training-videos) to assist in the training session. Study
- staff training may include review of the study CGM in real-time to make management decisions
- and how to review the data after an upload for retrospective review. Study staff will specifically
- identify how alarms are set using the app and the frequency that these alarms will repeat.
- For participants not using the Dexcom G6, the participants will be observed placing the sensor and
- will learn/review how to access the CGM trace via the Dexcom G6 commercial app (prior to the
- hotel session) and via the DiAs phone (during the hotel session). The participants will be asked to
- 429 perform fingerstick blood glucose measurements (if needed) in accordance with the labelling of
- 430 the study CGM device. An electronic copy of the CGM user's guide will be provided for these
- participants to read. The study team will be sure that the participants will leave the training session
- knowing how to properly use the CGM. The study team will be available for any questions.
- The study team will ask participants to share their data to the study Dexcom clinical account. This
- requires a one-time confirmation of data sharing between either the participant's personal Dexcom
- account or the study Dexcom account and the study clinical account. Participants are identified in
- 436 the study clinical account by their assigned participant number. The participant does not need to
- provide the study team with their own login information at any point in this process. The Dexcom
- dinical account allows the study team to remotely assess and download data as needed. Data
- sharing between the personal Dexcom account or study Dexcom account and the clinical account
- can be ended at any time by the participant.
- During Usual Care phase, participants will have the option of using their personal smartphone or
- receive a study smartphone to use in order to collect the data from the devices. They may also use
- their own Dexcom G6 or G7 CGM. If the participant elects to use a personal device, the Dexcom
- app will be downloaded to their phone in order to monitor the participant's CGM values and alerts
- in real-time may be used prior to initiating DiAs.

MiniNET 25-Oct-2024 

| 446 | 4.3 Blood Glucose Meter and Strips |
|---|---|
| 447 | 4.3.1 Equipment Description |
| 448<br>449 | A study glucometer will be provided to all participants to wear during the entire study to record any blood glucose levels measured during the study. |
| 450 | 4.3.2 Equipment Training |
| 451<br>452<br>453 | Participants will be advised to use the study glucometer when experiencing a low or high glucose values as defined in the Glycemic Treatment Guidelines. The Dexcom CGM will be calibrated, it needed, using the study glucometer and test strips in accordance with the manufacturer's labeling |
| 454<br>455<br>456<br>457 | If the study glucometer provides an app, the study team will request that the app be downloaded to the participant's personal phone. The app will permit continued visibility of blood glucose values to the participant and permit the study team to download the data without returning the glucometer at the end of the study. |
| 458 | 4.4 Ketone Meter and Strips |
| 459<br>460<br>461<br>462 | Blood ketone levels will be measured during the hotel and at-home portions of the study with either the Abbott Precision Xtra Meter or the Ketomojo Meters and ketone test strips in accordance with the manufacturer's labeling. Urine ketone strips may be provided to the participant for the athemed data collection period. The glucometer component of either ketone meters will not be used |
| 463 | 4.5 Study Devices Accountability Procedures |
| 464 | Device serial numbers will be recorded, and use of equipment will be tracked. |
| 465 | |

MiniNET\_25-Oct-2024 

# **Chapter 5: Randomization**

467 **VISIT 2** 

466

- Once eligibility is met and screening procedures are completed, the participant will proceed to
- Randomization. Participants will be randomized 1:1 to assess a 1-week usual care period before use of
- 470 the AIDANET system (Group A) or after use of the AIDANET system (Group B).
- 471 Participants who screen-fail or dropout will be replaced if it occurs prior to the Hotel Admission.
- 472 Randomization will occur via REDCap module.
- 473 GROUP A: Participants will complete one week at home usual care before the use of the
- 474 AIDANET system at the hotel admission.
- 475 **GROUP B**: Participants will complete one week at home usual care after the use of the AIDANET
- 476 system at the hotel admission.

MiniNET\_25-Oct-2024 

496

497

498

499

500

501

502

503

504

505

#### **Chapter 6: Usual Care Control Period** 477 478 6.1 Usual Care Control Period 479 VISIT 3 480 During the usual-care control period, participants will continue to use their personal insulin pump 481 in either manual or automated mode. The mode selected must be capable of downloading the data 482 and sharing it with the study team. Participants using Dexcom CGM will continue to use their 483 personal CGM or the study CGM and will share their CGM download data with the study team at 484 the completion of the Usual Care period. 485 All participants will be provided with a study glucometer to collect blood glucose values during 486 the study. This study team will download this glucometer at the conclusion of the study. 487 Participants will be instructed to follow their normal routine involving diet, exercise, and insulin 488 administration. 489 Any relevant contacts will be recorded on the CRF and summarized as appropriate (e.g. contact 490 that is not a scheduling or supplies issue will not be recorded). 491 **6.2 Pre-Hotel Check-In Visit** 492 VISIT 4 493 All participants will be contacted by the study team approximately 24-48 hours prior to the hotel 494 admission. The study team will verify the following information: 495

a. Inquire about any changes to the participant's medical history

- b. Study equipment (e.g., CGM) has been initiated. A new CGM sensor will be placed approximately 24-72 hours prior to the hotel session for proper warm-up.
- c. Verify with participant that the goal CGM reading at time of arrival is less than 200 mg/dL; this may require contact with the study physician prior to arrival on the day of the study visit.
- d. Participants will be encouraged to complete the INSPIRE and Technology Acceptance surveys prior to the hotel admission but no later than the initiation of the study equipment at the hotel admission.

Should any concerns regarding medical history, pump information, or unforeseen issues arise, the admission will be cancelled for that participant at the discretion of the investigator.

MiniNET 25-Oct-2024 

# **Chapter 7: Supervised Hotel Fully Closed Loop Period**

#### 507 **VISIT 5**

506

#### **7.1 Hotel Session**

- The study will be performed for about 36 hours at a local hotel/rental. Participants will use the
- AIDANET system in the hotel setting from the afternoon/evening of Day 1 through discharge in
- 511 the morning of Day 3. They will then continue to use the system for the at-home period of the
- 512 study.

513

## 7.2 Qualifications and Role of the Staff

- There will be at least two study staff present at all times at the study site, at least one of whom will
- be clinical staff (e.g., nurse, physician, nurse practitioner, physician assistant). There will be a
- 516 physician at the hotel or nearby on call during the study at all times. In addition, at least one senior
- engineer will be on call during the entire hotel session. Participants will be remotely monitored by
- at least one study team member (maybe trained staff, nurse, physician, NP, or PA) using a web-
- based remote monitoring system that has been previously established for DiAs. The web-based
- 520 remote monitoring system will display real-time insulin delivery, CGM and other system
- information to allow for patient safety monitoring. In addition, study team members will be trained
- 522 in all protocol and Glycemic Treatment Guideline procedures. The closed-loop system will be
- 523 managed by the participant with study-staff supervision, particularly at the time of insulin boluses
- 524 (if needed). Glucagon for the emergency treatment of hypoglycemia will be available on-site.
- Participants will be instructed to bring their own rescue glucagon, though each site will also bring
- 526 emergency rescue glucagon to the study.

#### **7.3 Hotel Session Check-In**

- Participants will arrive at the hotel on the first day of the hotel session. The study team will perform
- 529 vital signs and inquire about any changes to the participant's medical history. Any changes to
- medical history will be communicated to the medical physician to ensure continued eligibility and
- 531 participation.
- The participant 's CGM reading, and ketone concentration will be recorded. In the event that the
- participant's CGM reading is not between 80-250 mg/dL or ketone concentration is ≥0.6 mmol/L
- prior to initiation of the FCL system, the study physician may recommend additional insulin dosing
- according to the participants' usual doses. Study physician may elect to cancel participant's
- participation in the hotel admission if concerned about their medical safety. This participant will
- 537 not be replaced.
- The participant's home insulin pump will be discontinued, and the study insulin pump will be
- initiated. The study team will ensure the proper function of the CGM and insulin pump. The CGM
- used in the study is FDA-approved for the non-adjunctive measurement of blood glucose (i.e., the

MiniNET 25-Oct-2024 

- 541 CGM reading can be used for insulin dosing decisions). The CGM readings will be the primary
- source of blood glucose values. There is no required protocol fingerstick blood glucose
- measurements other than at times of CGM calibration (if necessary) and if directed by the study
- 544 team. Fingerstick blood glucose measurements may be taken whenever participants experience
- symptoms, if the CGM glucose is suspected to be erroneous, or any time the participant would like
- to be reassured. Glycemic Treatment Guidelines to be used during the hotel admission are defined
- 547 in section 7.6.

## **7.4 Study Meals**

- Participants will eat approximately 3 freely chosen unannounced meals per day during the
- supervised hotel session. Study staff will record the time the meal was eaten so that analysis of the
- AIDANET algorithm's performance around the mealtime may be conducted. Participants will use
- their usual insulin:carbohydrate ratio at dinner on Day 2. No other meal announcement will occur
- during the hotel stay. Snacks with carbohydrates will not be allowed unless for the treatment of
- low blood sugars. Non-carbohydrate snacks may be allowed throughout the hotel session per
- 555 investigator discretion. Blood glucose levels will be followed via CGM with interventions for
- glucose extremes as per the Glycemic Treatment Guidelines.

#### **7.5 Hotel Session Activities**

- Participants will engage in a walk of approximately 30 minutes on Day 2 of the hotel stay.
- Participants must have a CGM value of at least 80 mg/dL in order to begin the walk. The timing
- of exercise will be recorded by study staff so that analysis of the AIDANET algorithm's
- performance around exercise may be conducted. Participants will already be wearing an exercise
- monitor as part of the study protocol.
- The walk will be terminated early with subjective symptoms such as shortness of breath, chest
- pain, dizziness, palpitations, or any such concerning symptoms reported by participants.
- Participants will stop their participation in the exercise portion of the study if reporting any
- concerning symptoms. Study physicians (or physician's assistants) will assess the participants for
- their need for additional care outside the study. If symptoms resolve entirely and there is no
- additional requirement for care outside the study, participants may then continue with the
- remainder of the study per investigator discretion.
- Participants will also be free to engage in additional low-intensity activity (i.e., walking) during
- 571 the hotel admission. Study staff will accompany participants if they leave the house/hotel.

## **7.6 Glycemic Treatment Guidelines**

- 573 Hypo- and Hyperglycemia occurring while using the AIDANET system will be managed per the
- 574 following protocol during both the hotel and at-home portions of the trial. Glycemic Treatment
- 575 Guidelines will be available for staff use during the study sessions and will be provided to
- participants for the at-home phase of the study.

MiniNET 25-Oct-2024 

## **7.6.1 Hypoglycemia**

- a. If CGM falls below 70 mg/dL at any time, confirm <70mg/dL CGM readings and potential hypoglycemia symptoms with a fingerstick blood glucose. If blood glucose confirms <70mg/dL CGM reading, hypoglycemia will be treated with oral glucose of approximately 5-15 g. Participants will be encouraged to wait 15 min prior to giving a second glucose treatment. These fingerstick checks will be performed during the hotel stay and during the home portion if the participant chooses to do so. During the hotel stay we will also recheck a fingerstick blood glucose before retreatment.
- b. If a participant experiences any symptoms of hypoglycemia (e.g., shakiness, dizziness, sweating, pallor, clumsiness, difficulty paying attention, or tingling around the mouth), then the participant should treat with oral glucose of 5-15 g. Participants will be encouraged to wait 15 min prior to giving a second glucose treatment. During the hotel portion of the study, a fingerstick blood glucose will be assessed before such treatment for symptoms and before any re-treatment.
- c. If a participant displays any signs of neuroglycopenia (e.g., lethargy, disorientation, confusion, or inappropriate behavior) or severe hypoglycemia (e.g., hypoglycemic seizure, loss of consciousness, inability to properly consume treatment) hypoglycemia will be treated with either oral glucose or glucagon. The patient will be discharged from the study. The participant should consult with a study physician to discuss next steps for broader evaluation of symptoms unrelated to hypoglycemia.

## 7.6.2 Hyperglycemia

If CGM value is >300 mg/dL for 2 hours or >400 mg/dL at any time, check fingerstick BG and ketone level every 60±15 minutes. If unexplained hyperglycemia, evaluate the integrity of the insulin site, consider changing the site and providing a correction bolus as recommended by the bolus calculator. If insulin is given subcutaneous injection rather than through the DiAs, closed-loop control should be suspended for up to four hours unless directed by a study clinician.

## 7.7 FCL Equipment Training

- **VISIT 6**
- Participants will receive training on at-home use of the study system, safety protocols, and at-home
- study contacts on the day of discharge. Study equipment training is described in section Chapter
- 608 4:.

## 7.8 Hotel Session Discharge

- Discharge will occur after breakfast on Day 3. After discharge, participants will proceed to the
- Remote Monitored At-Home Phase of the study.

MiniNET 25-Oct-2024 

# 7.9 Other Issues The participant will be instructed to notify study staff if they experience any issues with the study devices. During the hotel phase, staff will provide hands-on support and troubleshooting training

- devices. During the hotel phase, staff will provide hands-on support and troubleshooting training for any device issues. If subcutaneous insulin is needed, the participant will turn off closed-loop
- mode as instructed by study staff. During the at-home phase, participants will be instructed to
- 617 mode as instructed by study starr. During the at-nome phase, participants will be instructed to contact the staff on-call in the event of subcutaneous insulin need. If insulin is delivered by any
- 618 means other than the study pump, the participant will be instructed to turn off closed-loop mode
- for approximately four hours. This timeframe can be adjusted by the study physician.
- The participant will also be asked to alert the study clinical staff for technical issues with the
- Tandem research pump and/or the DiAs system, including use of the study pump and study CGM
- 622 (open loop mode) during periods of component disconnections or technical difficulties.
- Glucagon will be available at the hotel once the investigational system is in place. All participants
- will confirm that they have rescue glucagon available at home for the at-home phase.

MiniNET 25-Oct-2024 

# **Chapter 8: Remote Monitored At-Home Fully Closed Loop Period**

#### 626 **VISIT 7**

625

## **8.1 At Home Participant Plan**

- Upon discharge on day 3 of the hotel period, participants will begin a 7 day/6-night Remote
- Monitored At-Home stage of the study. Participants will continue to wear the FCL research system
- as initiated during the hotel period. Participants will be instructed to eat approximately 3 freely
- chosen meals per day without announcing them to the system. The exception is that on 2 separate
- days participants will 1) announce all food intake (triggering an immediate BPS dose) and 2) use
- 633 their usual insulin-to-carbohydrate ratio for all food ingestion. Participants will be instructed to
- participate in their usual level of physical activity. Participants will complete the study after lunch
- on overall study day 9 (Day 7 of the home portion), at which point they will return to use of their
- usual diabetes care.
- Participants in Group A will complete the study after this 1-week FCL data collection period.
- Participants in Group B will then begin the Usual Care control period for data comparison (see
- 639 section 6.1).

## **8.2 Remote Monitoring**

- All participants will continue to be remote monitored during the At-Home period of the study
- using the connection between DiAs and Diabetes Web Monitoring (DWM) platform at UVA.
- Study staff may review the AID system data on the DWM platform as needed; in addition, at each
- site, a licensed medical provider (MD, PA, NP, RN, CDCES) will receive the following automated
- alerts from the DWM (automated notification system, ANS):
- 646 1. CGM > 300 mg/dL for 1 hour.
- 2. CGM < 70 mg/dL for 20 minutes.
- 648 3. CGM < 55 mg/dL at any point.
- 4. No sensor data for > 1 hour.
- The provider on call will contact study participants (e.g., call, text, or video chat) and/or their
- companion for any of the above CGM alerts which are not resolved within a timely manner.
- Participants will be asked to manage glycemic extremes per the hyper- hypoglycemia safety
- 653 protocol.
- 654 Contact (e.g., phone, text, email, etc.) with the study team will occur as needed. Any relevant
- contacts will be recorded on the CRF and summarized as appropriate (e.g. contact that is not a
- scheduling or supplies issue will not be recorded).

## **8.3 Questionnaires**

All participants will complete the INSPIRE and Technology Acceptance survey:

MiniNET 25-Oct-2024 

659

660

661 8.4 Post-Study Check-In 662 VISIT 8 663 Approximately 24-48 hours after the hotel session, the study team will contact the participant via 664 phone/email/text/video to: 665 • Ask about any changes to the participant's medical history and medication. Review any hypoglycemic events that are less than 60 mg/dL. 666 667 • Review any hyperglycemic events that are more than 300 mg/dL. • Verify that questions have been answered. The study physician or designee will be 668 669 available for any questions related to insulin adjustments/parameters. 670 The study team may contact the participant for issues related to data collection and equipment 671 issues. 672 **8.5** Early Termination Visit (If Applicable) Participants will be asked to attend the Post-Study Check-In Visit (visit 8) in the event of a 673 withdrawal or early termination. 674 675 8.6 Unscheduled Visits 676 Participants may have unscheduled visits during the study period if required for additional device training or other unanticipated needs per the study investigator discretion. 677

• Prior to initiating the study equipment at the hotel admission

At the conclusion of the one week of At-Home FCL data collection.

MiniNET 25-Oct-2024 

678

# **Chapter 9: Medical Monitor Safety Review**

The Medical Monitor will review compiled safety data at the conclusion of the trial. In addition, the Medical Monitor will review all DKA and severe hypoglycemia irrespective of relatedness to study device use, and all serious events (including UADEs) related to study device use at the time of occurrence. The Medical Monitor also will be informed of any Adverse Device Effects (ADE) not meeting criteria for a UADE if the Study PI requests the Medical Monitor review. The Medical Monitor can request modifications to the study protocol or suspension or stoppage of the study if deemed necessary based on the totality of safety data available.

MiniNET\_25-Oct-2024 

# 686 Chapter 10: Testing Procedures

## 10.1 Laboratory and Point of Care Testing

688 **10.1.1 HbA1c** 

687

698

716

- A blood sample (either capillary or venous draw) will be obtained at screening to obtain a baseline
- Hemoglobin A1c level. A blood test obtained within 4 weeks prior to enrollment may be used.
- HbA1c level may be measured by the study team using the DCA2000, a comparable point of care
- device, at time of screening. Labs may be obtained at a local laboratory (e.g., LabCorp, Quest)
- 693 convenient to the participant.

## 694 **10.1.2 Pregnancy Test**

- A serum or urine pregnancy test will be required for women of childbearing potential at in person
- of visit and admission. Test must be negative to participate in the study.

## 697 **10.2 Questionnaires**

#### 10.2.1 Demographic Data Survey

- Research in diabetes technology has revealed significant disparities in minoritized population's
- representation in clinical trials and access to devices that improve diabetes outcomes. Collection
- of detailed demographic data regarding participants in technology trials has become essential. This
- includes data on race/ethnicity, income levels and insurance status, as well as education and other
- variables that describe the study population.
- The Demographic Data Survey will be electronically administered once eligibility has been met.
- 705 The below information will be gathered for all participants.
- 706 a. Age
- 707 b. Gender
- 708 c. Race
- d. Ethnicity
- e. Martial status
- 711 f. Level of education
- g. Employment status
- 713 h. Household income
- 714 i. Health insurance status
- 715 j. Monthly insulin costs and co-payments

## 10.2.2 INSPIRE Questionnaire

- 717 The self-administered INSPIRE (INsulin Dosing Systems: Perceptions, Ideas, Reflections and
- Expectations) questionnaires have been developed to determine the psychosocial impact of AID

MiniNET 25-Oct-2024 
| 720 | with T1D, as well as parents/caregivers of youth with T1D, and partners of adults with T1D. |
|---|---|
| 721<br>722 | The questionnaire will be administered at the onset of hotel admission and at the conclusion of the study. |
| 723 | 10.2.3 Technology Expectations Survey |
| 724<br>725<br>726 | Participants will complete a Technology Expectation/Acceptance Survey which includes questions about attitudes, feelings, and behaviors related to the technology used in this study. AID Benefits and Burdens Scale Survey |
| 727<br>728 | The questionnaire will be administered prior to or at the onset of hotel admission and at the conclusion of the study. |

MiniNET\_25-Oct-2024 

734

739

746

755

# 29 Chapter 11: Risks Associated with the Clinical Trial

## 730 11.1 Potential Risks and Benefits of the Investigational Device

- Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are
- handled to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a
- risk in participants with type 1 diabetes and participants will be monitored for these symptoms.

### 11.1.1 Venipuncture Risks

- A hollow needle/plastic tube will be placed in the arm for taking blood samples. Blood draws can
- cause some common reactions like pain, bruising, or redness at the sampling site. Less common
- reactions include bleeding from the sampling site, formation of a small blood clot or swelling of
- 738 the vein and surrounding tissues, and fainting.

## 11.1.2 Fingerstick Risks

- About 1 drop of blood will be removed by fingerstick for measuring blood sugars and sometimes
- HbA1c or other tests. This is a standard method used to obtain blood for routine hospital laboratory
- 742 tests. Pain is common at the time of lancing. In about 1 in 10 cases, a small amount of bleeding
- under the skin will produce a bruise. A small scar may persist for several weeks. The risk of local
- infection is less than 1 in 1000. This should not be a significant contributor to risks in this study
- as finger sticks are part of the usual care for people with diabetes.

## 11.1.3 Subcutaneous Catheter Risks (CGM)

- Participants using the CGM will be at minimal risk for developing a local skin infection at the site
- of the sensor needle placement. If a needle is left under the skin for more than 24 hours, it is
- possible to get an infection where it goes into the skin, with swelling, redness and pain. There may
- be bleeding where the catheter is put in and bleeding under the skin causes a bruise (1 in 10 risk).
- 751 Study staff should verbally alert the participant that on rare occasions, the CGM may break and
- leave a small portion of the sensor under the skin that may cause redness, swelling, or pain at the
- 753 insertion site. The participant should be further instructed to notify the study coordinator
- 754 immediately if this occurs.

### 11.1.4 Risks of Hypoglycemia

- As with any person having type 1 diabetes and using insulin, there is always a risk of having low
- blood sugar (hypoglycemia). The frequency of hypoglycemia should be no more and possibly less
- 758 than it would be as part of daily living. Symptoms of hypoglycemia can include sweating,
- 759 jitteriness, and not feeling well. Just as at home, there is the possibility of fainting or seizures
- 760 (convulsions) and that for a few days the participant may not be as aware of symptoms of
- hypoglycemia. A CGM functioning poorly and significantly over-reading glucose values could
- 762 lead to inappropriate insulin delivery.

MiniNET 25-Oct-2024 

### 11.1.5 Risks of Hyperglycemia

Hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an extended period or if the pump or infusion set is not working properly. A CGM functioning poorly and significantly under-reading glucose values could lead to inappropriate suspension of insulin delivery.

#### 11.1.6 Risks of Device Reuse

- Participant will be informed that FDA or relevant national authorities have approved the insulin pump, CGM, glucometer and ketone meter for individual use and that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis B) may be spread through the use of multiple users.
- 773 The study CGM system is labelled for single patient use only. The sensor (the component of the system that enters the skin) will be individual use only. The transmitter and receiver may be reused during the study after the study team cleans the device using a hospital-approved cleaning
- procedure. The transmitter is attached to the sensor but does not enter the skin and the receiver, if
- used, is a handheld device.
- 778 CGM cleaning instructions are provided in the Dexcom G4 Platinum (Professional) Cleaning and
- 779 Disinfection manual (current edition) and a similar approach will be applied for the CGMs used in
- 780 this study.
- 781 The study insulin pumps are labelled for single patient use. During the study, this device may be
- reused after the study team cleans the device with a hospital-approved cleaning procedure. All
- infusion set equipment will be single patient use only (infusion set insertion kits, tubing, cartridges
- 784 etc.)

789

763

764

765766

767

768

769

770

771

772

- 785 The study-provided blood glucose meter will be returned to the study participant at the conclusion
- of the study after the study team has confirmed data collection. The study team will use cleaning
- procedures if it is necessary to be in physical contact with the equipment to download the device.
- 788 The study team will clean the ketone meter per manufacturer directions.

#### 11.1.7 Device Cleaning Instructions

- Members of the study team will clean the study equipment after use as noted in these instructions.
- 791 CGM cleaning instructions are provided in the Dexcom G4 PLATINUM (Professional) Cleaning
- and Disinfection manual (current edition). The transmitter should be cleaned with Clorox
- 793 Healthcare® Bleach Germicidal Cleaner or any disinfectant product in a spray bottle containing a
- bleach solution of 6500 parts per million with the EPA registration number 56392-7. The
- 795 transmitter will be submerged in this solution and then placed on an absorbent wipe or clean
- surface. Two sprays will be dispensed from the Clorox cleaner onto each side of the transmitter.
- 797 A nylon brush will be used to scrub the transmitter on all sides for 30 seconds. The transmitter

MiniNET 25-Oct-2024 

- 798 will be placed in the Clorox Cleaner solution for one minute. The transmitter is then rinsed under 799 flowing tap water for ten seconds. The transmitter will then be disinfected using a disinfectant product with EPA registration number 56392-7 using similar procedures as the cleaning process. 800 801 Per the pump manufacturer, the insulin pump will be cleaned with a damp lint-free cloth. Use of 802 household or industrial cleaners, solvents, bleach, scouring pads, chemicals, or sharp instruments 803 are prohibited. The pump should never be submerged in water. If needed, use only a very mild 804 detergent, such as a bit of liquid soap with warm water. A soft towel will be used to dry the pump. 805 The glucometer is cleaned and disinfected with two separate Super Sani-Cloths (EPA number 806 9480-4). The entire surface will be cleaned, making sure the surface stays wet for 2 minutes. This 807 step is repeated with a clean cloth for disinfecting the device. 808 The Precision Xtra User's Guide suggests that healthcare professionals use 10% bleach, 70% 809 alcohol or 10% ammonia to clean the device. 810 Equipment that touches intact skin will be cleaned with ethyl or isopropyl alcohol (70-90%), quaternary ammonium germicidal detergent (i.e. Cavicide, EPA number 46781) or household 811 812 bleach. The contact time on the surface depends on the method used to clean the equipment. 813 Cavicide requires three minutes on the surface of the equipment. Clorox Germicidal Bleach Wipes 814 require two minutes on the equipment. The surface should remain wet (i.e. slightly damp) with the 815 disinfectant to be considered effective though not wet enough to leave drops of liquid. 816 In the event a manufacturer updates cleaning procedures for their device, the study team will 817 adhere to the most current recommendations. 818 There is the risk of blood sampling collection and contamination from sampling techniques. Hand 819 washing with either soap & water or waterless hand sanitizer will be used prior to caring for the 820 study subject. Gloves will be worn during blood sample collection and processing. Medical personnel will continue to practice hygiene for the subject's protection (i.e. hand washing, 821 822 changing gloves frequently, disposing needles properly). Gloves will be removed, and hands 823 washed or sanitized prior to leaving and upon return to the subject's room. Soiled linen will be
  - 11.1.8 Hb1Ac Risk

changed to minimize the transfer of pathogenic organisms.

824

825

826

827

828

829

830

831

An NGSP Point of Care analyzer (i.e. DCA Vantage Analyzer) will be utilized at the research site to obtain the subject's HbA1c level.

#### 11.1.9 Other Risks

Some participants may develop skin irritation or allergic reactions to the adhesives used to secure the CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion. If these reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm,

MiniNET 25-Oct-2024 

- etc.) will be tried, sites will be rotated frequently, and a mild topical steroid cream or other
- medication may be required.
- Whenever the skin is broken there is the possibility of an infection. The CGM and pump infusion
- sites are inserted under the skin. It is possible that any part that is inserted under the skin may cause
- an infection. These occur very infrequently, but, if an infection was to occur, oral and/or topical
- antibiotics can be used. The risk of skin problems could be greater if you use a sensor for longer
- than it is supposed to be used. Therefore, participants will be carefully instructed about proper use
- 839 of the sensor.
- Data downloaded from the CGM, insulin pump, glucometer, and ketone meter will be collected
- 841 for the study as measures of diabetes self-management behaviors. Some people
- may be uncomfortable with the researchers' having such detailed information about their daily
- 843 diabetes habits.

844

848

860

### 11.1.10 Known Potential Benefits

- 845 It is anticipated that this protocol will yield increased knowledge about using an automated
- closed-loop system with anticipatory action to control glucose levels. The individual participant
- may not benefit from study participation.

#### 11.1.11 Risk Assessment

- Based on the facts that (1) adults and adolescents with diabetes experience mild hypoglycemia and
- 850 hyperglycemia frequently as a consequence of the disease and its management, (2) the study
- intervention involves periodic automated insulin dosing that may increase the likelihood of
- 852 hypoglycemia, and periodic automated attenuation of insulin delivery that may increase the
- likelihood of hyperglycemia, (3) mitigations are in place, and have been tested in prior studies
- using the investigational device system in the home setting, that limit the likelihood of excessive
- insulin dosing or prolonged withdrawal of insulin, and (4) rapid reversal of hypoglycemia and
- 856 hyperglycemia can be achieved, it is the assessment of the investigators that this protocol falls
- under DHHS 46.405 which is a minor increase over minimal risk. In addition, it is the belief of the
- 858 investigators that this study also presents prospects of direct benefit to the participants and general
- benefit to others with diabetes.

## 11.2 General Considerations

- The study is being conducted in compliance with the policies described in the study policies
- document, with the ethical principles that have their origin in the Declaration of Helsinki, with the
- protocol described herein, and with the standards of Good Clinical Practice (GCP).
- Whenever possible, data will be directly collected in electronic case report forms, which will be
- considered the source data.

MiniNET 25-Oct-2024 

866

867

868

The protocol is considered a significant risk device study, due to the fact that the closed loop system is experimental. Therefore, an investigational device exemption (IDE) from the U.S. Food and Drug Administration (FDA) is required to conduct the study.

MiniNET\_25-Oct-2024 

# Chapter 12: Adverse Events, Device Issues, and Stopping Rules

#### **12.1 Definitions**

## **12.1.1 Adverse Events (AE)**

- Any untoward medical occurrence in a study participant, irrespective of the relationship between
- the adverse event and the device(s) under investigation (section 12.2) for reportable adverse events
- for this protocol).

876

877

878

879

880

881

882 883

884

885

886 887

888

889

890

891

892

893

894

895896

897

898

899

900

901

Positive pregnancy test will not be considered an adverse event.

### 12.1.2 Serious Adverse Event (SAE)

- Any untoward medical occurrence that:
  - Results in death.
  - Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event).
  - Requires inpatient hospitalization or prolongation of existing hospitalization.
  - Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions (life threatening).
  - Is a congenital anomaly or birth defect.
  - Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the participant or may require medical/surgical intervention to prevent one of the outcomes listed above).

### 12.1.3 Unanticipated Adverse Device Effect (UADE)

Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of participants (21 CFR 812.3(s)).

### 12.1.4 Adverse Device Effect (ADE)

Any untoward medical occurrence in a study participant which the device may have caused or to which the device may have contributed.

#### 12.1.5 Device Complaints and Malfunctions

A device complication or complaint is something that happens to a device or related to device performance, whereas an adverse event happens to a participant. A device complaint may occur independently from an AE, or along with an AE. An AE may occur without a device complaint or there may be an AE related to a device complaint. A device malfunction is any failure of a device

MiniNET 25-Oct-2024 

to meet its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the labeling for the device. The intended performance of a device refers to the intended use for which the device is labeled or marketed. (21 CFR 803.3).

# 12.2 Reportable Events

For this protocol, a reportable adverse event includes any untoward medical occurrence that meets one of the following criteria:

- A serious adverse event as defined in section 12.1.2.
- An Adverse Device Effect as defined in section 12.1.4, unless excluded from reporting in section 12.7.
- An Adverse Event as defined in section 12.1.1 occurring in association with a study procedure.
- An AE as defined in section 12.1.1 which leads to discontinuation of a study device for 4 or more hours during the hotel phase and 12 or more hours during the at home phase.
- Hypoglycemia meeting the definition of severe hypoglycemia as defined in section 12.2.1
- Diabetic ketoacidosis (DKA) as defined in section 12.2.2 or in the absence of DKA, a hyperglycemic or ketosis event meeting the criteria defined below.

Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse events unless associated with an Adverse Device Effect. Skin reactions from sensor placement are only reportable if severe and/or required treatment.

### 12.2.1 Hypoglycemia Event

Hypoglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when the following definition for severe hypoglycemia is met:

- The event required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
- Impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma.
- If plasma glucose measurements are not available during such an event, neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.

### 12.2.2 Hyperglycemia Events/Diabetes Ketoacidosis

Hyperglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when one of the following four criteria is met:

MiniNET 25-Oct-2024 

940

941

942

943

944

945

947

948

949

950

955

961

962

963 964

965

966

967 968

969

970

971

- The event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and described below.
  - Evaluation or treatment was obtained at a health care provider facility for an acute event involving hyperglycemia or ketosis.
  - Blood ketone level  $\geq 1.5$  mmol/L and communication occurred with a health care provider at the time of the event.
  - Blood ketone level  $\geq$ 3.0 mmol/L, even if there was no communication with a health care provider.
- 946 Hyperglycemic events are classified as DKA if the following are present:
  - Symptoms such as polyuria, polydipsia, nausea, or vomiting.
  - Serum ketones ≥1.5 mmol/L or large/moderate urine ketones.
  - Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate <15.
  - Treatment provided in a health care facility.
- 951 All reportable Adverse Events—whether volunteered by the participant, discovered by study
- 952 personnel during questioning, or detected through physical examination, laboratory test, or other
- 953 means—will be reported on an adverse event form online. Each adverse event form is reviewed
- by the Medical Monitor to verify the coding and the reporting that is required.

## 12.3 Relationship of Adverse Event to Study Device

- The study investigator will review each adverse event and assess the relationship of any adverse
- event to be related or unrelated by determining if there is a reasonable possibility that the adverse
- event may have been caused by the study device.
- To ensure consistency of adverse event causality assessments, investigators should apply the following general guideline when determining whether an adverse event is related:
  - RELATED: There is a plausible temporal relationship between the onset of the adverse event and the study intervention, and the adverse event cannot be readily explained by the participant's clinical state, intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of response to the study intervention; and/or the adverse event abates or resolves upon discontinuation of the study intervention or dose reduction and, if applicable, reappears upon re-challenge.
  - UNRELATED: Evidence exists that the adverse event has an etiology other than the study intervention (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the adverse event has no plausible temporal relationship to study intervention.

# 12.4 Intensity of Adverse Event

The intensity of an adverse event will be rated on a three-point scale: (1) mild, (2) moderate, or (3) severe. It is emphasized that the term severe is a measure of intensity: thus, a severe adverse event

MiniNET 25-Oct-2024 

- 974 is not necessarily serious. For example, itching for several days may be rated as severe, but may 975 not be clinically serious.
  - MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities.
    - MODERATE: Usually causes a low level of inconvenience or concern to the participant and may interfere with daily activities but is usually ameliorated by simple therapeutic measures.
    - SEVERE: Interrupts a participant's usual daily activities and generally requires systemic drug therapy or other treatment.

### 12.5 Coding of Adverse Events

- Adverse events will be coded per standard categories (i.e., mild, moderate, severe). The Medical
- Monitor will review the investigator's assessment of causality and may agree or disagree. Both
- 986 the investigators and Medical Monitor's assessments will be recorded. The Medical Monitor will
- have the final say in determining the causality.
- Adverse events that continue after the participant's discontinuation or completion of the study will
- be followed until their medical outcome is determined or until no further change in the condition
- 990 is expected.

976

977

978

979

980

981

982

983

991

993

994

995

996

997 998

999

1000

1001

1002

1003

1004 1005

1006

1007

1008

1009

1010

#### 12.6 Outcome of Adverse Events

- The outcome of each reportable adverse event will be classified by the investigator as follows:
  - RECOVERED/RESOLVED The participant recovered from the AE/SAE without sequelae. Record the AE/SAE stop date.
  - RECOVERED/RESOLVED WITH SEQUELAE The event persisted and stabilized without change in the event anticipated. Record the AE/SAE stop date.
  - FATAL A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death.
  - NOT RECOVERED/NOT RESOLVED (ONGOING) An ongoing AE/SAE is defined as the event was ongoing with an undetermined outcome.
  - An ongoing outcome will require follow-up by the site in order to determine the final outcome of the AE/SAE.
  - The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date.
  - UNKNOWN An unknown outcome is defined as an inability to access the participant or the participant's records to determine the outcome (for example, a participant that was lost to follow-up).

MiniNET 25-Oct-2024 

- 1011 All clinically significant abnormalities of clinical laboratory measurements or adverse events
- 1012 occurring during the study and continuing at study termination should be followed by the
- participant's physician and evaluated with additional tests (if necessary) until diagnosis of the
- underlying cause, or resolution. Follow-up information should be recorded on source documents.
- 1015 If any reported adverse events are present when a participant completes the study, or if a participant
- 1016 is withdrawn from the study due to an adverse event, the participant will be contacted for re-
- evaluation within 2 weeks. If the adverse event has not been resolved, additional follow-up will be
- performed as appropriate. Every effort should be made by the Investigator or delegate to contact
- the participant until the adverse event has resolved or stabilized.

## 1020 **12.7 Reportable Device Issues**

- All UADEs, ADEs, device complaints, and device malfunctions will be reported irrespective of
- whether an adverse event occurred, except in the following circumstances.
- The following device issues are anticipated and will not be reported but will report as an Adverse
- 1024 Event if the criteria for AE reporting described above are met:
- Component disconnections

1026

1028

1029

1030

1031

1032

1033 1034

1035

1036

1037

1038

1039

1040 1041

1042

1043

1044 1045

1046 1047

1048

- CGM sensors lasting fewer than the number of days expected per CGM labeling
- CGM tape adherence issues
  - Pump infusion set occlusion not leading to ketosis
    - Battery lifespan deficiency due to inadequate charging or extensive wireless communication
    - Intermittent device component disconnections/communication failures not leading to system replacement
    - Device issues clearly addressed in the user guide manual that do not require additional troubleshooting
    - Skin reactions from CGM sensor placement or pump infusion set placement that do not meet criteria for AE reporting

### 12.8 Timing of Event Reporting

- UADEs must be reported within 10 working days to the FDA after the sponsor first receives notice of the adverse effect.
- Other reportable adverse events, device malfunctions (with or without an adverse event) and device complaints should be reported promptly, but there is no formal required reporting period.
- The IDE Sponsor will investigate the UADE and if indicated, report the results of the investigation to the IRBs, FDA, and Medical Monitor within 10 working days of the study team becoming aware of the UADE per 21CFR 812.46(b) (2).
- The Medical Monitor will determine if the UADE presents an unreasonable risk to participants. If so, the Medical Monitor must ensure that all investigations, or parts of investigations presenting that risk, are terminated as soon as possible but no later than

MiniNET 25-Oct-2024 

- 5 working days after the Medical Monitor makes this determination and no later than 1050 15 working days after first receipt notice of the UADE.
  - In the case of a device system component malfunction (e.g. pump, CGM, control algorithm), information will be forwarded to the responsible manufacturer by the study personnel.

## 12.9 Stopping Criteria

1051 1052

1053

1054

1055

1056

1057

1058 1059

1060

1061 1062

1063 1064

1065

1080

#### 12.9.1 Participant Discontinuation

A participant will be discontinued if any of the following occur:

- The investigator believes it is unsafe for the participant to continue the intervention. This could be due to the development of a new medical condition or worsening of an existing condition; or participant behavior contrary to the indications for use of the device that imposes on the participant's safety
- The participant requests that the treatment be stopped
- Two distinct episodes of DKA
- Two distinct severe hypoglycemia events as defined in section 12.2.1.
- Two events of any kind: severe hypoglycemia or DKA

## 12.9.2 Suspending/Stopping Overall Study

- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or severe hyperglycemia event (as defined in section 12.2.2), use of the study device system will be suspended while the problem is diagnosed.
- In the event that two distinct episodes of DKA or two distinct severe hypoglycemia events as defined in section 12.2.1 occur, the overall study would be suspended while the underlying conditions are determined.
- 1072 In addition, study activities could be similarly suspended if the manufacturer of any constituent
- study device requires stoppage of device use for safety reasons (e.g., product recall). The affected
- study activities may resume if the underlying problem can be corrected by a protocol or system
- modification that will not invalidate the results obtained prior to suspension. The study Medical
- Monitor will review all adverse events and adverse device events that are reported during the study
- and will review compiled safety data at periodic intervals. The Medical Monitor may request
- suspension of study activities or stoppage of the study if deemed necessary based on the totality
- of safety data available.

# 12.10 Independent Safety Oversight

- 1081 A Medical Monitor will review all DKA and severe hypoglycemia irrespective of relatedness to
- study device use, and all serious events (including UADEs) related to study device use at the time
- of occurrence. The Medical Monitor can request modifications to the study protocol or suspension
- or outright stoppage of the study if deemed necessary based on the totality of safety data available.

MiniNET 25-Oct-2024 

| Details regarding the Medical Monitor review will be documented in a separate Medical Monitor document. |
|---|
| 12.11 Definition of a Data Breach |
| A data breach is defined in the HITECH Act (43 USC 17932) as an unauthorized acquisition, |
| access, or use of protected health information (PHI) that compromises the security or privacy of |
| such information. |

MiniNET\_25-Oct-2024 

# 1091 Chapter 13: Miscellaneous Considerations

- 1092 13.1 Prohibited Medications, Treatments, and Procedures
- Participants using glulisine at the time of enrollment will be asked to contact their personal
- physician to change their prescribed personal insulin to lispro or aspart for the duration of the trial.
- The study devices (study insulin pump, study CGM) must be removed before Magnetic Resonance
- 1096 Imaging (MRI), Computed Tomography (CT) or diathermy treatment. Participants may continue
- in the trial after temporarily discontinuing use if requiring one of the treatments above.
- 1098 **13.2 Participant Withdrawal**
- Participation in the study is voluntary. Participant may withdraw at any time. For participants who
- do withdraw from the study, the study team will determine if their data will be used in analysis.
- 1101 **13.3 Confidentiality**
- For security and confidentiality purposes, subjects will be assigned an identifier that will be used
- instead of their name. Protected health information gathered for this study may be shared with the
- third-party collaborators. De-identified subject information may also be provided to collaborators
- involved in the study after the appropriate research agreement has been executed.
- 1106 **13.4 Lost to Follow Up**
- 1107 If a participant is lost to follow up and participant outcome cannot be determined, outcome
- classification will be the last known outcome/contact with the participant. A participant will be
- 1109 considered lost to follow-up after three attempted contacts that do not result in any communication
- from the participant. A certified letter may be sent as the fourth and final attempt to communicate
- 1111 with the participant.

MiniNET 25-Oct-2024 

1144

1145

# 1112 Chapter 14: Statistical Consideration

#### 1113 14.1 Design and Randomization 1114 The proposed work is a safety and feasibility study of the FCL system and is not intended to be powered to fully demonstrate efficacy of the system. The sample size of up to 6 participants per 1115 session at each site was selected based on previous experience of the feasible number of individuals 1116 1117 to supervise at one time under similar study conditions. 1118 14.1.1 Planned Analysis 1119 The primary outcome of interest will be the change in the mean CGM between the week of the Usual Care observational period and the week of AIDANET at-home. This study represents a 1120 small pilot study to assess the safety and efficacy of the small-version AIDANET system and is 1121 not formally powered. Nevertheless, the randomized crossover design will allow for analysis of 1122 period effects between Group A and Group B. Comparison between these groups will be made to 1123 1124 determine if a period effect can explain part of the benefit of the FCL system during the at-home 1125 period. a. Null Hypothesis: There is no difference in the mean CGM between the week of 1126 Usual Care observational period and the at-home FCL period. 1127 1128 b. Alternative Hypothesis: There is a difference in the mean CGM between the week of Usual Care observational period and the at-home FCL period. 1129 1130 Analysis will involve use of repeated measure ANOVA models to predict CGM average and TIR 1131 with the FCL status a fixed effect and baseline HbA1c and gender as covariates. 1132 Secondary outcomes: 1133 All secondary outcomes will be similarly analyzed. If an outcomes distribution is not suited for mixed model analysis (e.g., profound skewness, or large atom at boundary) we will perform paired 1134 Wilcoxon signed rank test (and loose the capacity to use covariate) to test difference in the median 1135 instead of the mean; this is expected for time below 70mg/dL, number of hypoglycemia, and 1136 1137 possibly time above 250mg/dL. 1138 We do not plan to correct for multiple comparisons. 1139 We do not expect substantial missing values in this supervised study, but if more than 3 participants 1140 have one or more missing admissions, we will consider switching from RANOVA to mixed model repeated measures. 1141 1142 14.2 Sample Size 1143 As an early exploratory study, the goal will be to complete 6 participants to provide data from a

MiniNET 25-Oct-2024 

variety of individuals. This number was chosen out of feasibility and not from a formal power

calculation. The total sample size of 6 participants was selected based on previous experience of

- the number of participants necessary to satisfy FDA requirements for a safety and feasibility study and move onto a larger out-patient efficacy study. While this sample size is thus a convenience
- sample, we may still determine the power to analyze each of the study hypotheses based on pilot
- 1149 trial data.

1150

1151

### 14.3 Outcome Measures

### 14.3.1 Primary Efficacy Endpoint

- The primary metric for analysis will be change in mean CGM between the second last 7 days week
- of the control Usual-Care period and the one-week Remote Monitored At-Home FCL period.

# 1154 **14.3.2 Secondary Outcomes**

- Glycemic Metrics will be obtained directly from CGM data and will include the standard metrics
- recommended by the international consensus on CGM including mean CGM, GMI derived from
- mean CGM, time in range 70-180 mg/dL, CGM standard deviation (StDev), CGM coefficient of
- variation (CV), CGM %<54 mg/dL, CGM %<70 mg/dL, CGM %>180 mg/dL, and CGM %>250
- 1159 mg/dL. For the Usual Care period, CGM data will be obtained from either the participant's
- personal CGM or a study provided CGM. Data for the control Usual-Care period will be analyzed
- by last available 7-day period. During the FCL period, CGM data will be obtained directly from
- the study device. As GMI is a linear transformation of mean CGM, this metric will have the same
- effect and will be presented as a primary outcome as well. All other glycemic metrics will be
- 1164 considered secondary outcome measures.
- Device-Use Metrics will include time in automation, total daily insulin dose, and number of
- boluses per day. During the Usual Care period, participants using an insulin pump will have their
- pump uploaded at the end of the period to capture their insulin delivery and bolus data. The FCL
- period, insulin use, and bolus data (if any) will be captured from the experimental device.
- Exercise Challenge Metrics will include the duration of exercise, approximate intensity of exercise
- (low, moderate, or high intensity), the % CGM<70 mg/dL, % CGM<54 mg/dL, and any episodes
- of SH (CGM<70mg/dL for more than 15 minutes with interruption, CGM≥70, of less than 15
- minutes or CHO treatment) during and 2 hours after the exercise challenges.
- 1173 Unannounced Meal Metrics during the supervised house/hotel FLC stage participants will be
- instructed to eat at least 3 meals per day. The time of completion for these meals will be recorded
- by study staff. The % CGM>250 mg/dL for the 4 hours after each meal will be recorded and
- specifically analyzed. Participants will be instructed to freely eat meals during the supervised at-
- home FCL stage but will not be required to record the timing of the meals for unannounced meals.
- Patient Reported Outcomes will include several surveys aiming to capture participant satisfaction
- 1179 with the FCL device and any changes in distress or burden of diabetes management. See
- 1180 APPENDIX for survey tools. These surveys will include:

MiniNET 25-Oct-2024 

| 1181<br>1182 | a. The INSPIRE Measures: A validated tool assessing the positive expectancies of AID systems for youth, adults, and parents and partners of people with diabetes. This tool |
|---|---|
| 1183 | has been specifically endorsed by the FDA for use with developing insulin-dosing |
| 1184<br>1185 | systems. b. Technology Expectations Surveys: A 25 question self-report measure of |
| 1186<br>1187 | expectations from advanced technologies and perceived impact of the technology on quality of life. Validated to age 13+ years. |
| 1188<br>1189 | These surveys will be administered at baseline and then at the end of the prior to or at the start of the 1-week supervised House/Hotel FCL period and at the end of the 1-week remote-monitored |
| 1190 | at-home FCL study |
| 1191 | 14.3.3 CGM Data Treatment |
| 1192<br>1193 | a. Saturated CGM values "High" and "Low" will be replaced by 401mg/dL and 39mg/dL respectively. |
| 1194 | b. Any CGM gaps shorter than 1 hour will be interpolated |
| 1195 | c. CGM data during recorded occlusion event will be removed from analysis as |
| 1196 | follows: any measurement less than 2h before or after the time of record will be |
| 1197 | removed. |
| 1198 | d. CGM data following a pump/DiAs communication interruption >1h by less than 2h |
| 1199 | will be removed |
| 1200 | 14.3.4 Outcome Computation Conditions |
| 1201<br>1202 | Outcomes will only be computed if at least 80% of the analysis window CGM measurements (after data treatment) are available. |
| 1203 | 14.4 Safety Analyses |
| 1204<br>1205<br>1206 | We will assess for the system's functionality, including the ability of the system to run its code without error (delivering insulin safely, as planned), as well as its ability to avoid low BG $<$ 70 mg/dL. |
| 1207 | 14.5 Baseline Descriptive Statistics |
| 1208 | Baseline demographic and clinical characteristics of the cohort of all randomized participants will |
| 1209<br>1210 | be summarized in a table using summary statistics appropriate to the distribution of each variable. Descriptive statistics will be displayed overall and by treatment group. |
| 1211 | Will include: |
| 1212 | a. Age |
| 1213 | b. HbA1c |
| 1214 | c. Gender |

MiniNET\_25-Oct-2024 

| 5 | d. Race/ethnicity |
|---|---|
| 6 | e. CGM use before enrollment |
| 7 | f. AID use before enrollment |
| 8 | g. Diabetes duration |
| 9 | h. BMI |
| 0 | i. Total Daily Insulin |
| 1 | 14.6 Device Issues |
| 2 | The following tabulations and analyses will be performed during time on the UVa AP systems to |
| 3 | assess device issues: |
| 4 | a. Device malfunctions requiring study team contact and other reported device issues |
| 5 | b. % time CGM data available |
| 6 | c. % time with closed loop control |

MiniNET\_25-Oct-2024 

# 1227 Chapter 15: Data Collection and Monitoring

### 1228 **15.1 Case Report Forms and Device Data**

- The study data are collected through a combination of case report forms (electronic and paper) and
- 1230 electronic device data files obtained from the software and individual hardware components.
- 1231 These electronic device files and electronic CRFs are considered the primary source
- 1232 documentation.
- 1233 When data are directly collected in electronic case report forms, this will be considered the source
- 1234 data. Records will be maintained in accordance with ICH E6 and institutional regulatory
- requirements for the protection of confidentiality of participants.

# 1236 **15.2 Study Records Retention**

- 1237 Study documents should be retained for a minimum of 2 years after the last approval of a marketing
- application in an ICH region and until there are no pending or contemplated marketing applications
- in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical
- development of the investigational product. These documents should be retained for a longer
- period, however, if required by local regulations. No records will be destroyed without the written
- 1242 consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the
- investigator when these documents no longer need to be retained.

#### 1244 **15.3 Protocol Deviations**

- 1245 A protocol deviation is any noncompliance with the clinical trial protocol, Good Clinical Practices
- 1246 (GCP), or procedure requirements. The noncompliance may be either on the part of the participant,
- the investigator, or the study site staff. As a result of deviations, corrective actions may be
- developed by the site and implemented as appropriate. Major deviations will be reported to the
- 1249 IRB-HSR within 7 calendar days of when the study team becomes aware of the event.

MiniNET 25-Oct-2024 

# **Chapter 16: Ethics/Protection of Human Participants**

#### **1251 16.1 Ethics Standard**

1255

1262

1263

1264

1265 1266

1267

1268

1269

1270

1271

1272

- The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21
- 1254 CFR Part 56, and/or the ICH E6.

### 16.2 Institutional Review Boards

- 1256 The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- form must be obtained before any participant is enrolled. Any amendment to the protocol will
- require review and approval by the IRB before the changes are implemented to the study. All
- 1260 changes to the consent form will be IRB approved; a determination will be made regarding whether
- previously consented participants need to be re-consented.

### **16.3 Informed Consent Process**

#### 16.3.1 Consent Procedures and Documentation

Informed consent is a process that is initiated prior to an individual's agreement to participate in the study and continues throughout the individual's study participation. The potential participant will be provided with a short overview of the study including its study goals, study procedures, and study timeline. If the potential participant remains interested, they will be asked permission to review inclusion/exclusion criteria to assess if they are eligible to participate in the study. If permission is granted, the study team will review the Inclusion/Exclusion criteria (section 3.4 and 3.5). If eligible, the study team member will provide a copy of the informed consent form (e.g., in person, email, fax, or mail) to the potential participant for their review. Potential participants may also elect to review the informed consent form prior to discussing pre-screening questions.

- The potential participant will be provided with ample time to read and review the consent form.
- 1274 After their review, the study team will discuss the study at length in a phone call/HIPAA compliant
- telecommunication method for consenting that is not face to face. All participants will receive
- verbal explanation in terms suited to their comprehension of the purposes, procedures, and
- potential risks of the study and of their rights as research participants. Extensive discussion of risks
- and possible benefits of participation will be provided. The potential participant will be given an
- opportunity to ask the study team questions or may speak directly with the study physician. The
- potential participant's understanding of the information presented in the process of consent will be
- assessed by asking open-ended questions.
- The consent form may be signed electronically for both in-person and telecommunication
- screening visits. Note: For potential participants who are not able to sign an electronic consent
- form, in-person, email, fax, or mail will be alternatives used to obtain a signed consent. A HIPAA

MiniNET 25-Oct-2024 

1303

compliant video conferencing tool (e.g., Zoom, WebEx) will be utilized during the consenting 1285 process of the telecommunication screening visit to facilitate the FDA Part 11 compliant process 1286 of verification of reviewing two forms of identification if signing electronically off site. 1287 Participants can download a PDF copy of the signed consent and automatically receive a PDF via 1288 email from REDCap after the form is completed. CRCs also could download, print, and mail a 1289 1290 paper copy for each participant. Study procedures may begin once the consent has been signed by the participant and a member of the study team. 1291 1292 The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study. 1293 1294 16.4 Participant and Data Confidentiality 1295 The IRB-HSR Post Approval Monitoring (PAM) auditors, representatives of the IRB, or device 1296 company supplying study product may inspect documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) for the 1297 participants in this study. 1298 1299 The study participant's contact information will be securely stored at the clinical site for internal 1300 use during the study. At the end of the study, all records will continue to be kept in a secure location 1301 for as long a period as dictated by local IRB and institutional regulations. The study data entry and 1302 study management systems used by research staff will be secured and password protected. At the

end of the study, all study databases will be archived at the UVA CDT.

MiniNET\_25-Oct-2024 

# 1304 Chapter 17: References

- 1305 1. Rogers MAM, Kim C, Banerjee T, Lee JM. Fluctuations in the incidence of type 1 diabetes in the 1306 United States from 2001 to 2015: a longitudinal study. BMC medicine. 2017;15(1):199.
- 2. Forlenza GP, Rewers M. The epidemic of type 1 diabetes: what is it telling us? Current opinion in endocrinology, diabetes, and obesity. 2011;18(4):248-51.
- 3. Committee ADAPP. 6. Glycemic Targets: Standards of Medical Care in Diabetes—2022. Diabetes Care. 2021;45(Supplement 1):S83-S96.
- 4. Committee ADAPP. 14. Children and Adolescents: Standards of Medical Care in Diabetes—2022.
   Diabetes Care. 2021;45(Supplement 1):S208-S31.
- Malik FS, Sauder KA, Isom S, Reboussin BA, Dabelea D, Lawrence JM, et al. Trends in Glycemic
   Control Among Youth and Young Adults With Diabetes: The SEARCH for Diabetes in Youth Study.
   Diabetes Care. 2022;45(2):285-94.
- 6. Sawyer A, Sobczak M, Forlenza GP, Alonso GT. Glycemic Control in Relation to Technology Use in a Single Center Cohort of Children With Type 1 Diabetes. Diabetes technology & therapeutics. 2022.
- 7. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. The Diabetes Control and Complications Trial Research Group. N Engl J Med. 1993;329(14):977-86.
- 1321 8. Lachin JM, Genuth S, Nathan DM, Zinman B, Rutledge BN. Effect of glycemic exposure on the risk of microvascular complications in the diabetes control and complications trial--revisited. Diabetes. 2008;57(4):995-1001.
- 9. Pop-Busui R, Herman WH, Feldman EL, Low PA, Martin CL, Cleary PA, et al. DCCT and EDIC studies in type 1 diabetes: lessons for diabetic neuropathy regarding metabolic memory and natural history. Current diabetes reports. 2010;10(4):276-82.
- 10. Jacobson AM, Braffett BH, Cleary PA, Gubitosi-Klug RA, Larkin ME. The long-term effects of type 1 diabetes treatment and complications on health-related quality of life: a 23-year follow-up of the Diabetes Control and Complications/Epidemiology of Diabetes Interventions and Complications cohort. Diabetes Care. 2013;36(10):3131-8.
- 1331 11. Nathan DM, Bayless M, Cleary P, Genuth S, Gubitosi-Klug R, Lachin JM, et al. Diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: advances and contributions. Diabetes. 2013;62(12):3976-86.
- 1334 12. Nathan DM. The diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: overview. Diabetes Care. 2014;37(1):9-16.
- 13. Berget C, Messer LH, Forlenza GP. A Clinical Overview of Insulin Pump Therapy for the Management of Diabetes: Past, Present, and Future of Intensive Therapy. Diabetes spectrum: a publication of the American Diabetes Association. 2019;32(3):194-204.
- 1339 14. Forlenza GP, Kushner T, Messer LH, Wadwa RP, Sankaranarayanan S. Factory-Calibrated Continuous
   1340 Glucose Monitoring: How and Why It Works, and the Dangers of Reuse Beyond Approved Duration
   1341 of Wear. Diabetes technology & therapeutics. 2019.
- 1342 15. Forlenza GP, Lal RA. Current Status and Emerging Options for Automated Insulin Delivery Systems.
  1343 Diabetes technology & therapeutics. 2022.

MiniNET 25-Oct-2024 

- 1344 16. Kowalski A. Pathway to artificial pancreas systems revisited: moving downstream. Diabetes Care. 2015;38(6):1036-43.
- 17. Kowalski AJ. Can we really close the loop and how soon? Accelerating the availability of an artificial pancreas: a roadmap to better diabetes outcomes. Diabetes technology & therapeutics. 2009;11 Suppl 1:S113-9.
- 1349 18. Ware J, Allen JM, Boughton CK, Wilinska ME, Hartnell S, Thankamony A, et al. Randomized Trial 1350 of Closed-Loop Control in Very Young Children with Type 1 Diabetes. N Engl J Med. 1351 2022;386(3):209-19.
- 1352 19. Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, et al. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019.
- 20. Breton MD, Kanapka LG, Beck RW, Ekhlaspour L, Forlenza GP, Cengiz E, et al. A Randomized Trial of Closed-Loop Control in Children with Type 1 Diabetes. N Engl J Med. 2020;383(9):836-45.
- 1356
   21. McAuley SA, Trawley S, Vogrin S, Ward GM, Fourlanos S, A. Grills C, et al. Closed-Loop Insulin
   1357
   Delivery Versus Sensor-Augmented Pump Therapy in Older Adults With Type 1 Diabetes (ORACL):
   A Randomized, Crossover Trial. Diabetes Care. 2021:dc211667.
- 22. Collyns OJ, Meier RA, Betts ZL, Chan DSH, Frampton C, Frewen CM, et al. Improved Glycemic
   Outcomes With Medtronic MiniMed Advanced Hybrid Closed-Loop Delivery: Results From a
   Randomized Crossover Trial Comparing Automated Insulin Delivery With Predictive Low Glucose
   Suspend in People With Type 1 Diabetes. Diabetes Care. 2021;44(4):969-75.
- 23. McAuley SA, Lee MH, Paldus B, Vogrin S, de Bock MI, Abraham MB, et al. Six Months of Hybrid
   Closed-Loop Versus Manual Insulin Delivery With Fingerprick Blood Glucose Monitoring in Adults
   With Type 1 Diabetes: A Randomized, Controlled Trial. Diabetes Care. 2020;43(12):3024-33.
- 24. Messer LH, Berget C, Pyle L, Vigers T, Cobry E, Driscoll KA, et al. Real-World Use of a New Hybrid
   Closed Loop Improves Glycemic Control in Youth with Type 1 Diabetes. Diabetes technology &
   therapeutics. 2021.
- Da Silva J, Lepore G, Battelino T, Arrieta A, Castañeda J, Grosman B, et al. Real-world Performance
   of the MiniMed<sup>TM</sup> 780G System: First Report of Outcomes from 4'120 Users. Diabetes technology &
   therapeutics. 2021.
- 26. Breton MD, Kovatchev BP. One Year Real-World Use of the Control-IQ Advanced Hybrid Closed Loop Technology. Diabetes technology & therapeutics. 2021.
- 27. Berget C, Akturk HK, Messer LH, Vigers T, Pyle L, Snell-Bergeon J, et al. Real world performance of hybrid closed loop in youth, young adults, adults and older adults with type 1 diabetes: Identifying a clinical target for hybrid closed loop use. Diabetes, obesity & metabolism. 2021.
- 28. Amadou C, Franc S, Benhamou PY, Lablanche S, Huneker E, Charpentier G, et al. Diabeloop DBLG1
   Closed-Loop System Enables Patients With Type 1 Diabetes to Significantly Improve Their Glycemic
   Control in Real-Life Situations Without Serious Adverse Events: 6-Month Follow-up. Diabetes Care.
   2021;44(3):844-6.
- 1381
   29. Stone MP, Agrawal P, Chen X, Liu M, Shin J, Cordero TL, et al. Retrospective Analysis of 3-Month
   Real-World Glucose Data After the MiniMed 670G System Commercial Launch. Diabetes technology
   & therapeutics. 2018;20(10):689-92.
- 30. Forlenza GP, Breton MD, Kovatchev B. Candidate Selection for Hybrid Closed Loop Systems.

  Diabetes technology & therapeutics. 2021.

MiniNET 25-Oct-2024 

1388

1389

| 1386 | 31. Fredette ME, Zonfrillo MR, Park S, Quintos JB, Gruppuso PA, Topor LS. Self-reported insulin pump |
|---|---|
| 1387 | prescribing practices in pediatric type 1 diabetes. Pediatr Diabetes. 2021. |

32. Pauley ME, Berget C, Messer LH, Forlenza GP. Barriers to Uptake of Insulin Technologies and Novel Solutions. Med Devices (Auckl). 2021;14:339-54.

MiniNET\_25-Oct-2024 